CLINICAL TRIAL: NCT00144157
Title: An Open-Label Study of Nevirapine Plus Combivir® (ZDV+3TC) Treatment in Women Who Have Previously Received a Nevirapine Regimen for the Prevention of Mother to Child Transmission (pMTCT) of HIV-1.
Brief Title: Open Label Study of NVP+CBV Treatment in Women Who Have Received sdNVP for the pMTCT of HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1414
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine
Drug: 3TC

SUMMARY:
To determine the response to treatment with NVP, ZDV and 3TC in HIV positive women, who previously received NVP for the prevention of mother to child transmission.

DETAILED DESCRIPTION:
An open-label, single arm, multicentre study to determine the virologic and immunologic responsiveness of women, who previously received a regimen of nevirapine for the prevention of MTCT, to a regimen of nevirapine and ZDV+3TC treatment. As well as to evaluate the proportion of patients who fail this treatment at 24 and 48 weeks, and to evaluate the resistance profile of HIV isolates from patients who fail nevirapine and ZDV+3TC treatment.

Study Hypothesis:

When a drug leading to selection of a resistant viral population is withdrawn the original wildtype virus, over time, becomes the predominant virus again. However, low frequency (below level of detection) of drug resistant viral sub-populations may be retained which could mean that the drug resistant variant might reappear rapidly should the same drug be reintroduced as part of combination therapy at a later stage.Therefore this study is proposed to evaluate whether there is an impact of single dose nevirapine for the prevention of MTCT on the subsequent response to a standard HAART regimen that contains nevirapine.

Comparison(s):

trial 1100.1090

ELIGIBILITY:
INCLUSION CRITERIA

* HIV-1-infected non-pregnant women who received a nevirapine regimen, for the prevention of mother to child transmission, at least 12 months previously.
* Women of child-bearing potential must have a negative urine pregnancy test at the screening visit and ensure double barrier methods of contraception, which by definition will in all cases include the use of condoms, throughout the study period.
* CD4 cell count < 350 cells/mm3 and viral load HIV-1 RNA > 20,000 c/mL or any symptomatic individual (WHO stage 3) or the presence of any AIDS defining criteria.
* Documented HIV-1 positive status by a licensed HIV-1 ELISA test.

EXCLUSION CRITERIA

* Women who are pregnant or breastfeeding.
* Women with prior exposure to antiretroviral therapy, other than a nevirapine regimen for the prevention of mother to child transmission at least 12 months previously.
* Subjects who in the investigator's opinion are unlikely to complete the 48 week study period or unlikely to comply with the dosing schedule and protocol evaluations.
* Patients with a Karnofsky performance status score < 70.
* Subjects who fail to meet the HIV treatment criteria (CD4 and viral load) indicated above.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2003-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07

PRIMARY OUTCOMES:
The proportion of patients who fail to suppress viral load to 400c/mL or maintain a viral load 400 c/mL at 24 and 48 weeks. The mean change in HIV RNA measurement by 24 weeks.

SECONDARY OUTCOMES:
What type of resistance that develops Immunologic response to treatment Treatment safety Time to treatment and/or virologic failure 5.How many achieve viral loads<50c/mL

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. South Africa (Pty.) Ltd.
Locations (3):
- South Africa (3):
  - Boehringer Ingelheim Investigational Site, Capetown
  - Boehringer Ingelheim Investigational Site, Parow
  - Boehringer Ingelheim Investigational Site, Soweto